CLINICAL TRIAL: NCT06872294
Title: Research of Predictive Factors of in Vitro Fertilization (IVF) Outcome in Women Affected by Autoimmune Disorders: From Biological Markers to Artificial Intelligence
Brief Title: Research of Predictive Factors of in Vitro Fertilization (IVF) Outcome AI-IVF Study
Acronym: AI-IVF
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Università degli Studi di Pavia (Unknown)
Responsible Party: Principal Investigator, Claudia Omes, Principal investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: AI-IVF
Record Dates: First submitted 2025-02-18; First posted 2025-03-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with a positive autoimmune panel: Women undergoing ART procedures with a positive autoimmune panel
- patients with a negative autoimmune panel: Women undergoing ART procedures with a negative autoimmune panel

SUMMARY:
Infertility is the failure to achieve a clinical pregnancy after 12 months or more of regular unprotected intercourse, while subfertility means a delay in achieving pregnancy. Several factors can contribute to these conditions, such as autoimmune diseases like systemic thyroid and celiac diseases, rheumatoid arthritis, systemic lupus erythematosus, and endometriosis. Some of them may overlap, sharing a common immunological milieu.

In this scenario, medically ART can help women carry on pregnancies if they are in stable disease remission and receive adequate treatment. However, the number of oocytes that can be ovulated under stimulation is highly variable, so the outcome of any IVF is linked to many factors, not only biological but also connected to the mean success rate of the fertility center.

For these reasons, the need to find methods for identifying the best gametes and embryos to guarantee a successful pregnancy is becoming pressing. AI can be essential to develop prediction models for pregnancy outcomes for patients undergoing ART treatments.

AI currently represents a modern way to obtain algorithms from a set of observable data that could help clinical decisions

ELIGIBILITY:
Inclusion Criteria:

* Women with age below 43 years old
* IVF cycle with fresh semen sample that could be used
* progressive motile spermatozoa expected count of minimum 1 million following density gradient purification on the day of oocyte pick up

Exclusion Criteria:

* Women with uterine abnormalities
* Women with chromosomal and genetic abnormalities
* Positivity to serological test (HCV, HBV, HIV, VDRL-TPHA)

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing ART procedures (n= 200, ) at SSD Ostetricia e Ginecologia 2 - PMA of Fondazione IRCCS Policlinico San Matteo, Pavia (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Predictive algorithm creation | through study completion, an average of 2 years
  Probability to achieve a pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Omes, PhD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (1):
- SSD Ostetricia e Ginecologia 2 - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No